CLINICAL TRIAL: NCT02473367
Title: A Study to Evaluate the Influence of Metal Cation-Containing Antacids on MK-0518 Pharmacokinetics in HIV-Infected Subjects on a Stable Raltegravir-Containing Regimen
Brief Title: The Effect of Antacids on the Pharmacokinetics (PK) of Raltegravir in Human Immunodeficiency Virus (HIV)-Infected Participants (MK-0518-824)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0518-824
Record Dates: First submitted 2015-06-12; First posted 2015-06-16 (Estimated); Results first posted 2016-09-01 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2018-07

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Raltegravir Pre- and 4 Period Sequence (Experimental): Starting five days prior to Period 1 participants will be treated with 1200 mg raltegravir, once daily for five days. In Period 1 participants will be treated with 1200 raltegravir alone; this is followed by Period 2 where participants will be treated with 1200 mg raltegravir and TUMS concomitantly; this is followed by Period 3 where participants will be treated with 1200 mg raltegravir and 12 hours later with Leader Antacid; followed by Period 4 where participants will be treated with 1200 mg raltegravir and 12 hours later with TUMS. The wait between Periods is 2-7 days.
  Interventions: Drug: Raltegravir 1200 mg; Drug: TUMS; Drug: Leader Antacid

INTERVENTIONS:
Drug: Raltegravir 1200 mg — Two tablets of 600 mg raltegravir administered orally, once daily, over 5 days of Pre-treatment, and once at the start of Periods 1-4.
Drug: TUMS — Three tablets of TUMS Ultra Strength (US) 1000, taken orally, concomitantly with raltegravir in Period 2, and 12 hours after raltegravir in Period 4
Drug: Leader Antacid — 20 mL Leader Antacid Maximum Strength (MS) taken orally 12 hours after raltegravir, in Period 3

SUMMARY:
In order to define the safe windows for co-dosing of metal-cation antacids with once daily administered raltegravir, this study will evaluate the effect of both calcium carbonate and magnesium/aluminum hydroxide antacids on the pharmacokinetics of raltegravir, due to dosage of 1200 mg raltegravir in HIV-infected participants already taking 400 mg raltegravir twice daily as part of their HIV treatment regimen.

ELIGIBILITY:
Inclusion Criteria:

* Is HIV positive
* Is on a stable raltegravir-containing (400 mg every 12hr) antiretroviral (ARV) regimen for at least 1 month prior to study entry, with no changes, including dose adjustments; and agrees to maintain their current ARV therapy throughout the study.
* Be male, or a non-pregnant and non-breast feeding female at least 18 years of age at the pre-trial (screening)
* Has a Body Mass Index (BMI) =< 32 kg/m^2

Exclusion Criteria:

* Has a history of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary or major neurological (including stroke and chronic seizures) abnormalities or diseases (excluding HIV)
* Has a history of gastric bypass surgery
* Has a history of cancer (malignancy)
* Has a history of chronic diarrhea within approximately 3 months prior to the pre-trial visit
* Has a history of significant multiple and/or severe allergies (e.g. food, drug, latex allergy), or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food
* Has had major surgery, donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks prior to the pre-trial visit
* Has participated in another investigational trial within 4 weeks prior to the pre-trial visit
* Is currently taking rifampin or atazanavir or is unable to refrain from the use of 1) any proton pump inhibitor from two weeks prior to the study through the completion of Period 4, and 2) any H2-blockers, over-the-counter antacids, calcium supplements or multivitamins from one week prior to the study through the completion of Period 4
* Consumes greater than 3 glasses of alcoholic beverages or distilled spirits per day
* Consumes greater than 6 servings of coffee, tea, cola, energy-drinks, or other caffeinated beverages per day
* Is currently a regular user (including "recreational use") of any illicit drugs or has a history of drug (including alcohol) abuse within approximately 6 months of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-06-23 (Actual); Primary Completion 2015-08-29 (Actual); Study Completion 2015-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Krishna R, East L, Larson P, Valiathan C, Butterfield K, Teng Y, Hernandez-Illas M. Effect of metal-cation antacids on the pharmacokinetics of 1200 mg raltegravir. J Pharm Pharmacol. 2016 Nov;68(11):1359-1365. doi: 10.1111/jphp.12632. Epub 2016 Sep 27. PMID 27671833

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Males or females, at least 18 years of age, with HIV infection were enrolled in this trial.
Pre-assignment Details: Starting five days prior to Period 1 participants were treated with 1200 mg raltegravir (MK-0518), once daily for five days.
Groups:
- Four Period Fixed Sequence: All participants entered the first of four treatment periods. Period 1: 1200 mg raltegravir alone; followed by Period 2: 1200 mg raltegravir and TUMS Ultra Strength (US) 1000 taken orally concomitantly; followed by Period 3: 1200 mg raltegravir and 12 hours later with 20 mL Leader Antacid Maximum Strength (MS) taken orally; followed by Period 4: 1200 mg raltegravir and 12 hours later with three tablets of TUMS US 1000 taken orally. There was a maximum 7-day wait between each period where participants were treated once daily with 1200 mg raltegravir.
Period: Period 1
Arm/Group | Four Period Fixed Sequence
Started | 20
Completed | 20
Not Completed | 0
Period: Wait 1
Arm/Group | Four Period Fixed Sequence
Started | 20
Completed | 19
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Period 2
Arm/Group | Four Period Fixed Sequence
Started | 19
Completed | 19
Not Completed | 0
Period: Wait 2
Arm/Group | Four Period Fixed Sequence
Started | 19
Completed | 19
Not Completed | 0
Period: Period 3
Arm/Group | Four Period Fixed Sequence
Started | 19
Completed | 19
Not Completed | 0
Period: Wait 3
Arm/Group | Four Period Fixed Sequence
Started | 19
Completed | 19
Not Completed | 0
Period: Period 4
Arm/Group | Four Period Fixed Sequence
Started | 19
Completed | 18
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- All Enrolled Participants: All participants who enrolled in the study
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.8 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 18

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration Time Curve From Time 0 to 24 Hrs (AUC 0-24hr) of Raltegravir Following Once Daily Administration of Raltegravir
Description: In Period 1 participants were treated with 1200 mg raltegravir alone; followed by Period 2 where participants were treated with 1200 mg raltegravir and three tablets of TUMS Ultra Strength (US) 1000 taken orally concomitantly; followed by Period 3 where participants were treated with 1200 mg raltegravir and 12 hours later with 20 mL Leader Antacid Maximum Strength (MS) taken orally; followed by Period 4 where participants were treated with 1200 mg raltegravir and 12 hours later with three tablets of TUMS US 1000 taken orally. The wait between Periods was a maximum of 7 days, during which participants were treated with 1200 mg raltegravir once daily. To determine the plasma concentration of raltegravir, blood samples were collected from pre-dose up to 24 hours post-dose, and analysis of variance (ANOVA) modeling was performed on natural log-transformed values to derive geometric least-squares means.
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose
Population: Per-Protocol: Participants who complied with the protocol sufficiently to ensure that generated data would reflect the effects of treatment, according to the underlying scientific model.
Measure: Least Squares Mean (95% Confidence Interval); unit: hr*µM
Groups:
- Period 1: Raltegravir Only: 1200 mg raltegravir, once at the start of Period 1
- Period 2: Raltegravir + TUMS Concomitantly: 1200 mg raltegravir and three tablets of TUMS US 1000 concomitantly once at the start of Period 2
- Period 3: Raltegravir + 12 Hrs Leader Antacid: 1200 mg raltegravir once at the start of Period 3, and 12 hours later with 20 mL Leader Antacid MS
- Period 4: Raltegravir + 12 Hrs TUMS: 1200 mg raltegravir once at the start of Period 4, and 12 hours later with 3 tablets of TUMS US 1000
Arm/Group | Period 1: Raltegravir Only | Period 2: Raltegravir + TUMS Concomitantly | Period 3: Raltegravir + 12 Hrs Leader Antacid | Period 4: Raltegravir + 12 Hrs TUMS
Number analyzed (Participants) | 20 | 19 | 19 | 19
hr*µM | 53.7 [44.2 to 65.2] | 14.8 [12.4 to 17.7] | 46.3 [36.0 to 59.6] | 48.5 [39.0 to 60.3]
Statistical Analysis 1: Comparison: Period 1: Raltegravir Only vs Period 2: Raltegravir + TUMS Concomitantly; Test type: Superiority or Other; Geom. least-squares mean ratio (GLSMR) = 0.28, 90% CI 2-sided [0.24 to 0.32] — Raltegravir+TUMS/Raltegravir only
Statistical Analysis 2: Comparison: Period 1: Raltegravir Only vs Period 3: Raltegravir + 12 Hrs Leader Antacid; Test type: Superiority or Other; GLSMR = 0.86, 90% CI 2-sided [0.73 to 1.03] — Raltegravir+12 Hrs Leader Antacid/Raltegravir only
Statistical Analysis 3: Comparison: Period 1: Raltegravir Only vs Period 4: Raltegravir + 12 Hrs TUMS; Test type: Superiority or Other; GLSMR = 0.90, 90% CI 2-sided [0.80 to 1.03] — Raltegravir+12 Hrs TUMS/Raltegravir only

2. Primary Outcome: Maximum Plasma Concentration (Cmax) of Raltegravir Following Once Daily Administration of Raltegravir
Description: In Period 1 participants were treated with 1200 mg raltegravir alone; followed by Period 2 where participants were treated with 1200 mg raltegravir and three tablets of TUMS US 1000 taken orally concomitantly; followed by Period 3 where participants were treated with 1200 mg raltegravir and 12 hours later with 20 mL Leader Antacid MS taken orally; followed by Period 4 where participants were treated with 1200 mg raltegravir and 12 hours later with three tablets of TUMS US 1000 taken orally. The wait between Periods was a maximum of 7 days, during which participants were treated with 1200 mg raltegravir once daily. To determine the plasma concentration of raltegravir, blood samples were collected from pre-dose up to 24 hours post-dose, and ANOVA modeling was performed on natural log-transformed values to derive geometric least-squares means.
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: nM
Arm/Group | Period 1: Raltegravir Only | Period 2: Raltegravir + TUMS Concomitantly | Period 3: Raltegravir + 12 Hrs Leader Antacid | Period 4: Raltegravir + 12 Hrs TUMS
Number analyzed (Participants) | 20 | 19 | 19 | 19
nM | 20000 [16500 to 24300] | 5240 [4230 to 6490] | 17300 [12800 to 23300] | 19500 [15900 to 24000]
Statistical Analysis 1: Comparison: Period 1: Raltegravir Only vs Period 2: Raltegravir + TUMS Concomitantly; Test type: Superiority or Other; GLSMR = 0.26, 90% CI 2-sided [0.21 to 0.32] — Raltegravir+TUMS/Raltegravir only
Statistical Analysis 2: Comparison: Period 1: Raltegravir Only vs Period 3: Raltegravir + 12 Hrs Leader Antacid; Test type: Superiority or Other; GLSMR = 0.86, 90% CI 2-sided [0.65 to 1.15] — Raltegravir+12 Hrs Leader Antacid/Raltegravir only
Statistical Analysis 3: Comparison: Period 1: Raltegravir Only vs Period 4: Raltegravir + 12 Hrs TUMS; Test type: Superiority or Other; GLSMR = 0.98, 90% CI 2-sided [0.81 to 1.17] — Raltegravir+12 Hrs TUMS/Raltegravir only

3. Primary Outcome: Plasma Concentration at 24 Hrs Post-dose (C24hr) of Raltegravir Following Once Daily Administration of Raltegravir
Description: In Period 1 participants were treated with 1200 mg raltegravir alone; followed by Period 2 where participants were treated with 1200 mg raltegravir and three tablets of TUMS US 1000 taken orally concomitantly; followed by Period 3 where participants were treated with 1200 mg raltegravir and 12 hours later with 20 mL Leader Antacid MS taken orally; followed by Period 4 where participants were treated with 1200 mg raltegravir and 12 hours later with three tablets of TUMS US 1000 taken orally. The wait between Periods was a maximum of 7 days, during which participants were treated with 1200 mg raltegravir once daily. To determine the plasma concentration of raltegravir, blood samples were collected at 24 hours post-dose, and ANOVA modeling was performed on natural log-transformed values to derive geometric least-squares means.
Time Frame: 24 hours post-dose
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: nM
Arm/Group | Period 1: Raltegravir Only | Period 2: Raltegravir + TUMS Concomitantly | Period 3: Raltegravir + 12 Hrs Leader Antacid | Period 4: Raltegravir + 12 Hrs TUMS
Number analyzed (Participants) | 20 | 19 | 19 | 19
nM | 75.6 [55.3 to 103] | 39.6 [29.9 to 52.5] | 32.0 [23.7 to 43.2] | 32.4 [24.6 to 42.6]
Statistical Analysis 1: Comparison: Period 1: Raltegravir Only vs Period 2: Raltegravir + TUMS Concomitantly; Test type: Superiority or Other; GLSMR = 0.52, 90% CI 2-sided [0.45 to 0.61] — Raltegravir+TUMS/Raltegravir only
Statistical Analysis 2: Comparison: Period 1: Raltegravir Only vs Period 3: Raltegravir + 12 Hrs Leader Antacid; Test type: Superiority or Other; GLSMR = 0.42, 90% CI 2-sided [0.34 to 0.52] — Raltegravir+12 Hrs Leader Antacid/Raltegravir only
Statistical Analysis 3: Comparison: Period 1: Raltegravir Only vs Period 4: Raltegravir + 12 Hrs TUMS; Test type: Superiority or Other; GLSMR = 0.43, 90% CI 2-sided [0.36 to 0.51] — Raltegravir+12 Hrs TUMS/Raltegravir only

ADVERSE EVENTS:
Time Frame: Periods 1-3: up to 24 hours after treatment with raltegravir; Period 4: up to 14 days after treatment with raltegravir
Description: Participants who received at least one dose of raltegravir
Arm/Group | Period 1: Raltegravir Only | Period 2: Raltegravir + TUMS Concomitantly | Period 3: Raltegravir + 12 Hrs Leader Antacid | Period 4: Raltegravir + 12 Hrs TUMS
Serious Adverse Events (participants affected / at risk) | 0/20 | 1/19 | 0/19 | 1/19
Other Adverse Events (participants affected / at risk) | 9/20 | 4/19 | 5/19 | 5/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1: Raltegravir Only (N=20) | Period 2: Raltegravir + TUMS Concomitantly (N=19) | Period 3: Raltegravir + 12 Hrs Leader Antacid (N=19) | Period 4: Raltegravir + 12 Hrs TUMS (N=19)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1: Raltegravir Only (N=20) | Period 2: Raltegravir + TUMS Concomitantly (N=19) | Period 3: Raltegravir + 12 Hrs Leader Antacid (N=19) | Period 4: Raltegravir + 12 Hrs TUMS (N=19)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 2 (2) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.